CLINICAL TRIAL: NCT06378619
Title: Machine Learning Analysis Of The Tapping Test And The Archimedean Spiral For The Differential Diagnosis Of Essential Tremor And Parkinson's Disease.
Brief Title: Tapping Test and the Archimedean Spiral for the Differential Diagnosis of Tremor. Machine Learning Approach
Acronym: MATSEP
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-50
Record Dates: First submitted 2024-04-15; First posted 2024-04-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Tremor; Essential Tremor; Parkinson Disease
Keywords: Tremor; Essential Tremor; Parkinson Disease; Diagnosis, Differential; Machine Learning
MeSH Terms: conditions — Tremor; Essential Tremor; Parkinson Disease; Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Essential Tremor: Tris group will include 55 participants affected by essential tremor
  Interventions: Diagnostic Test: Tapping Test; Diagnostic Test: Archimedes Spiral
- Parkinson Disease: Tris group will include 55 participants affected by Parkinson Disease
  Interventions: Diagnostic Test: Tapping Test; Diagnostic Test: Archimedes Spiral

INTERVENTIONS:
Diagnostic Test: Tapping Test — For the administration of the tapping test, a computer application installed on a Tablet will be used. The test will be administered up to 3 times, with a 15-minute interval between each administration. Each tapping test trial will last 15 seconds. At the beginning of the session, the patient will perform 2 practice attempts.
Diagnostic Test: Archimedes Spiral — For the administration of the Archimedean spiral, a computer application installed on a Tablet will be used. The Tablet screen will display a drawing of the spiral, serving as a reference for the participant. The test will be administered up to 3 times, with a 15-minute interval between each administration. At the beginning of the session, the patient will perform 2 practice attempts.

SUMMARY:
In clinical practice, it is sometimes difficult to establish whether a patient's tremor is due to Parkinson's disease or essential tremor. The distinction is crucial as the health implications differ significantly between the two conditions. Therefore, the present study aims to develop a diagnostic method based on machine learning techniques to help differentiate whether a patient's tremor is due to one condition or the other. To achieve this, 110 patients with tremor, correctly diagnosed with either Parkinson's disease or essential tremor, will participate. They will undergo two diagnostic tests (tapping test and Archimedean spiral) to capture data that can be processed using machine learning techniques.

ELIGIBILITY:
Inclusion Criteria:

* Possibility to collaborate in the necessary evaluations.
* Follow-up in the specialized consultation of Movement Disorders at the Neurology Service of Hospital Sant Camil-Consorci Sanitari Alt Penedes i Garraf.
* Legal capacity to provide informed consent.
* Signature of informed consent for study inclusion, either by the participant themselves or by their legal representative.
* Participant with criteria from Group 1 or 2:

Group 1:

* Confirmed diagnosis of tremor due to Parkinson's disease, clinically established, based on the diagnostic criteria of the Movement Disorders Society, and additionally:
* Tremor associated with bradykinesia of any duration.
* Confirmatory clinical diagnosis of tremor due to Parkinson's disease (stages 1 to 2 of Hoehn and Yahr) by the neurologist responsible for the participant's follow-up.

Group 2:

* Confirmed diagnosis of essential tremor, based on the criteria of the Movement Disorders Society, and additionally:
* Positional tremor plus kinetic and/or resting tremor with follow-up in outpatient neurology consultations for at least 3 years without a change in diagnosis.
* Absence of bradykinesia.

Exclusion Criteria:

* Patients undergoing treatment with antipsychotics or antidepressants.
* Patients with Parkinson's disease and dyskinesias.
* Patients undergoing treatment with dopaminergic agonists or primidone.
* Tremor of such severity that it prevents continuous tracing, at the investigator's discretion.
* Cognitive or affective pathology that limits the ability to collaborate with the study procedures.
* Participation in another clinical study involving an intervention, procedure, or visit frequency that is incompatible with the present study.
* Participants diagnosed with any of the following conditions:

Alcoholism of sufficient intensity to influence handwriting or cause neuropathy, at the investigator's discretion. Peripheral neuropathy of any cause. Dystonias. Previous stroke.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be contacted based on the patient registry with follow-up in the neurology clinic of the study center.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | through study completion, an average of 1 year
  Proportion of participants with confirmed Parkinson's disease for whom the machine learning-based diagnostic algorithm yields a 'positive' result.
Specificity | through study completion, an average of 1 year
  Proportion of participants with confirmed essential tremor for whom the machine learning-based diagnostic algorithm yields a 'negative' result.

SECONDARY OUTCOMES:
Reliability | through study completion, an average of 1 year
  The reliability of the diagnostic algorithm will be evaluated based on the repeatability of the classification result (positive or negative) among the different tests conducted on the same patient

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Camacho, MD, Principal Investigator — Consorsi Sanitari Alt Penedes i Garraf
Locations (1):
- Hospital Sant Camil-Consorci Sanitari Alt'Pènedes i Garraf, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.